CLINICAL TRIAL: NCT06741670
Title: Determination of the Effects of Three Different Methods in Reducing Pain During Heel Blood Collection; Breastfeeding, Vibration, and Breastfeeding+Vibration: A Randomized Controlled Study
Brief Title: Effects of Three Different Methods in Reducing Pain During Heel Blood Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Selda Ateş Beşirik, Principal Investigator, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GO 2024/412
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Newborn; Pain Management; Breastfeeding; Vibration; Wounds, Penetrating; Needlestick Injuries
Keywords: Newborn; Pain; Breastfeeding; Vibration; Heel Blood Collection
MeSH Terms: conditions — Agnosia; Breast Feeding; Wounds, Penetrating; Needlestick Injuries; Pain | interventions — Lactation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Prospective, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Breastfeeding Group (Experimental): Breastfeeding was applied to the infants in this group before and during the heel lance procedure.
  Interventions: Behavioral: Breastfeeding
- Vibration Group (Experimental): Vibration was applied to the infants in this group before and during the heel lance procedure.
  Interventions: Device: Vibration
- Breastfeeding+Vibration Group (Experimental): Breastfeeding+Vibration was applied to the infants in this group before and during the heel lance procedure.
  Interventions: Other: Breastfeeding+Vibration
- Control Group (No Intervention): In this group, infants received routine heel blood collection procedure.

INTERVENTIONS:
Behavioral: Breastfeeding — The routine practice of the Breastfeeding Group is to place the infants in their mother's arms and start breastfeeding 1 minute before the procedure. Then, the nurse will take the heel blood.
  Arms: Breastfeeding Group
Device: Vibration — The vibration device was placed on the infant's left extremity in the mid/lateral region just below the knee where the sural nerve passes. The device was secured to the extremity with a gauze bandage. The infants in the Vibration Group will be placed in their mother's arms and vibration will be applied 30 seconds before the routine application, and vibration will be applied during the 10-second waiting phase while the nurse performs the heel prick blood collection procedure.
  Arms: Vibration Group
Other: Breastfeeding+Vibration — The vibration device was placed on the infant's left extremity in the mid/lateral region just below the knee where the sural nerve passes. The device was secured to the extremity with a gauze bandage.
  The routine practice for the Breastfeeding+Vibration Group babies will be started by holding them in their mother's arms and breastfeeding will be started 1 minute before the application. At the same time, vibration will be applied 30 seconds before the application and vibration will be applied in a 10-second waiting phase while the nurse performs the heel prick procedure.
  Arms: Breastfeeding+Vibration Group

SUMMARY:
This prospective study is planned as a randomized controlled study with the purpose of determining the effect of Breastfeeding, Vibration, and Breastfeeding+Vibration on pain levels during heel blood collection on healthy term newborn's.

DETAILED DESCRIPTION:
Among the non-pharmacological methods frequently used to reduce the effects of invasive interventions on the newborn; Practices such as reducing environmental stimuli, individualized developmental care, music therapy, breast milk, pacifier giving, sucrose, non-nutritive sucking, oral sucrose, kangaroo care, facilitated tucking position, and sweet solutions, massage and touching, positioning, nesting, kangaroo care, fetal positioning are included.

This study is a prospective, randomized and controlled trial. In this study aim, the effect of Breastfeeding, Vibration, and Breastfeeding+Vibration during heel blood collection on the pain levels in healthy term newborn's will be examined.

Sample of the study consisted of a total of 192 newborns who met the sample selection criteria and were selected via randomization method. Newborns were divided into four groups; Breastfeeding group (n=48), Vibration group (n=48), Breastfeeding+Vibration group (n=48), and Control group (n=48).

Data were collected using the Infant-family Information Form and NIPS-Neonatal Infant Pain Scale. Data collection All blood sampling was performed in a quiet nursery room between 09:00 AM and 11:00 AM, 1-2 hours after breastfeeding, the normal time when infants undergo heel stick for routine blood collection for metabolic screening. Blood collection was performed in a standardized manner by the same nurse who has a minimum of 5 years' experience in the performance heel stick and had no conflict of interest. A pediatrician made the clinical decision for heel stick.

Before the procedure, the newborns were kept in a quiet room far away from the cries of other babies. The infants' diapers were changed before procedure. For the heel stick procedure, the antiseptic solution (70% alcohol), heel stick method, heel region for sampling (the outer right side of the ball), needle (21-G needle), and environmental factors such as heat, light, and noise were all standardized. The whole procedure was video-recorded until three minutes after the procedure.

At the beginning of the study, the parents of the newborns were informed about the aim and content of the research, and parental approval was obtained. Neonatal and family demographics were collected using self-report information forms, which included medical history, mother's gestational age, neonatal age, sex, birth weight, duration of sampling, total crying time, processing time, and the time from the start of the first cry to the first crying during the process.

All blood sampling in the study was performed for clinical purposes, such as newborn metabolic screening tests, which were taken on the second to third days following birth. The standard protocol for blood sampling involved swabbing the heel with a small gauze pad with disinfectant, lancing the heel, and then gently squeezing the heel intermittently until the amount of blood required for clinical use was collected.

All procedures performed in the experimental and control groups were video recorded by the researcher from the beginning of the procedure. After the procedure the newborns' pain levels and crying duration were evaluated using the video recordings. Assessment of pain was conducted independently by the investigator and the nurse using NIPS. At the same time, the newborns' total procedural crying time, the duration of the procedure, and the first calming time were recorded. The total crying time of the newborns was measured from the start of crying due to heel stick to the complete cessation of crying. The time of the procedure was measured from the beginning to the end of the heel stick procedure. The calming time was measured from the time of the first cry to the first calming time.

ELIGIBILITY:
Inclusion Criteria:

* Parents who volunteered and gave consent to participate in the research
* Full term neonates (38-42 weeks of gestation)
* Underwent heel stick blood drawing for routine metabolic screening,
* Aged 2 to 4 days
* Passed the hearing screening
* Birth weight between 2500-4400 grams
* Parents who know how to read, write and speak Turkish.

Exclusion Criteria:

* Parents with any mental problems
* Infants with any chronic disease and congenital anomalies.

Ages: 2 Days to 4 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
NIPS (Neonatal Infant Pain Scale) | average 5 minutes) during the heel blood collection procedures (1 minute before the heel lance procedure (T-1 minute), during the procedure (T+0 second), and 2 minutes (T+2 minutes)]
  It was developed by Lawrence et al. in 1993 to evaluate interventional pain in newborns (Lawrence et al, 1993). Its Turkish adaptation was made by Akdovan and Yıldırım in 1999. NIPS is an assessment tool that focuses on six behavioral responses of newborns: facial expressions, crying, breathing, arm movements, leg movements, and arousal. A score between 0 and 7 is obtained from the scale, and as the score obtained from the scale increases, the pain of newborns also increases. In the Turkish adaptation study of the scale, the Cronbach's alpha value was calculated as 0.83 before the procedure, 0.83 during the procedure and 0.86 after the procedure.

SECONDARY OUTCOMES:
Crying times | [Time Frame: during the heel blood collection procedures (average 5 minutes)]
  Duration of crying were recorded.
Processing time | [Time Frame: during the heel blood collection procedures (average 5 minutes)]
  Duration of heel blood collection procedure were recorded.
The time to first calming | [Time Frame: Procedure (The calming time was measured from the time of the first cry to the first calming time.) (average 5 minutes)]
  The calming time was measured from the time of the first cry to the first calming time.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Ateş Beşirik, Principal Investigator — Burdur Mehmet Akif Ersoy University
Locations (1):
- Burdur Mehmet Akif Ersoy University, Burdur, Bucak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this study, after deidentification, will be shared with researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code